CLINICAL TRIAL: NCT04531280
Title: Hospital-Level Care at Home for Acutely Ill Adults in Rural and Ultra-Rural Settings: Proof of Concept
Brief Title: Rural Home Hospital: Proof of Concept
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Rx Foundation (Other)
Responsible Party: Principal Investigator, David Levine, Dr. David Levine MD, MPH, MA, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020P000708
Record Dates: First submitted 2020-08-02; First posted 2020-08-28 (Actual); Results first posted 2025-01-30 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2024-12

CONDITIONS: Infection; Heart Failure; Chronic Obstructive Pulmonary Disease; Asthma; Gout Flare; Chronic Kidney Diseases; Hypertensive Urgency; Atrial Fibrillation Rapid; Anticoagulants; Increased
Keywords: home hospital; hospital at home; hospital in the home
MeSH Terms: conditions — Infections; Heart Failure; Pulmonary Disease, Chronic Obstructive; Asthma; Renal Insufficiency, Chronic; Hypertensive Crisis | interventions — Home Care Services, Hospital-Based

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Home hospital care (Experimental): Patients receive hospital-level care in their home, as a substitute to traditional hospital care
  Interventions: Other: Home hospital care

INTERVENTIONS:
Other: Home hospital care — Patients receive hospital-level care in their home.

SUMMARY:
This study examines the implications of providing hospital-level care in rural homes.

DETAILED DESCRIPTION:
Home hospital care is hospital-level care at home for acutely ill patients. In multiple publications mostly in urban environments, home hospital care delivered cost-effective, high-quality, excellent experience care with similar quality and safety as traditional hospital care. Most home hospital models deliver care in urban environments, not in rural environments.

To further improve the model, the investigators propose to determine the feasibility of home hospital care in a rural home setting through a proof-of-concept approach.

ELIGIBILITY:
Patient clinical inclusion Criteria:

* >=18 years old
* Any infectious process (e.g., pneumonia, diverticulitis, cellulitis, complicated urinary tract infection)
* Heart failure exacerbation
* Asthma and chronic obstructive pulmonary disease exacerbation
* Atrial fibrillation with rapid ventricular response
* Diabetes and its complications
* Venous thromboembolism: This includes a patient who requires therapeutic anticoagulation and concomitant monitoring (thus requiring inpatient status)
* Gout exacerbation
* Chronic kidney disease with volume overload
* Hypertensive urgency
* End of life / desires only medical management: Regarding a patient who desires only medical management, this includes a patient who requires acute care for symptom management but declines any surgical intervention. This may include a patient who is about to transition to hospice care, for example, but still has the functional capacity to meet our criteria below. Under these circumstances, we would make sure that various contingencies, including possible transition to hospice care or hospital readmission, are completely understood by patients and caregivers as applicable.

Patient social inclusion criteria:

* Lives in rural or ultra-rural area (see definitions in Appendix) that can be served by one of our RHH clinicians.
* Has capacity to consent to study
* Can identify a potential caregiver who agrees to stay with patient for first 24 hours of admission. Caregiver must be competent to call care team if a problem is evident to her/him. After 24 hours, this caregiver should be available for as-needed spot checks on the patient: This criterion maybe waived for highly competent patients at the patient and clinician's discretion.

Patient caregiver inclusion criteria: (not required for patient participation):

* Age >= 18 years old
* Has capacity to consent to study
* Lives with or nearby to patient

Clinician inclusion criteria:

-Any member of the rural home hospital (RHH) clinical team (MD, RN, paramedic, NP) who will be participating in the screening and recruitment of patients for the rural home hospital intervention and/or providing care to rural patients that enroll in the intervention.

Patient Clinical Exclusion Criteria:

* Acute delirium, as determined by the Confusion Assessment Method
* Cannot establish peripheral access (or access requires ultrasound guidance, unless ultrasound guidance is available)
* Secondary condition: active non-melanoma/prostate cancer, end-stage renal disease, acute myocardial infarction, acute cerebral vascular accident, acute hemorrhage
* Primary diagnosis requires controlled substances
* Cannot independently ambulate to bedside commode
* As deemed by on-call MD, patient likely to require any of the following procedures that have not already occurred: computed tomography, magnetic resonance imaging, endoscopic procedure, blood transfusion, cardiac stress test, or surgery
* For pneumonia: Most recent CURB65 > 3: new confusion, BUN > 19mg/dL, respiratory rate>=30/min, systolic blood pressure<90mmHg, Age>=65 (<14% 30-day mortality); Most recent SMRTCO > 2: systolic blood pressure < 90mmHg (2pts), multilobar CXR involvement (1pt), respiratory rate >= 30/min, heart rate >= 125, new confusion, oxygen saturation <= 90% (<10% chance of intensive respiratory or vasopressor support); Absence of clear infiltrate on imaging; Cavitary lesion on imaging; Pulmonary effusion of unknown etiology; O2 saturation < 90% despite 5L O2
* For heart failure: Has a left ventricular assist device; GWTG-HF17 (>10% in-hospital mortality) or ADHERE18 (high risk or intermediate risk 1)*; Severe pulmonary hypertension
* For complicated urinary tract infection: Absence of pyuria; Most recent qSOFA > 1 (SBP≤100 mmHg, RR≥22, GCS<15 [any AMS]) (if sepsis, >10% mortality)
* For other infection: Most recent qSOFA > 1 (SBP≤100 mmHg, RR≥22, GCS<15 [any AMS]) (if sepsis, >10% mortality)
* For COPD: BAP-65 score > 3 (BUN>25, altered mental status, HR>109, age>65) (<13% chance in-hospital mortality): exercise caution
* For asthma: Peak expiratory flow < 50% of normal: exercise caution
* For diabetes and its complications: Requires IV insulin
* For hypertensive urgency: Systolic blood pressure > 190 mmHg; Evidence of end-organ damage; for example, acute kidney injury, focal neurologic deficits, myocardial infarction
* For atrial fibrillation with rapid ventricular response: Likely to require cardioversion; New atrial fibrillation with rapid ventricular response; Unstable blood pressure, respiratory rate, or oxygenation; Despite IV beta and/or calcium channel blockade in the emergency department, HR remains > 125 and SBP remains different than baseline; Less than 1 hour of time has elapsed with HR < 125 and SBP similar or higher than baseline
* For patients with end-stage renal disease on peritoneal dialysis: Peritoneal catheter malfunction; Requires temporary hemodialysis
* Home hospital census is full (maximum 3 patients at any time)

  * GWTG-HF: AHA Get with the Guidelines: SBP, BUN, Na, Age, HR, Black race, COPD ADHERE: Acute decompensated heart failure national registry: BUN, creatinine, SBP

Patient social exclusion criteria:

* Non-english speaking
* Undomiciled
* No working heat (October-April), no working air conditioning if forecast > 80°F (June-September), or no running water
* On methadone requiring daily pickup of medication
* in police custody
* Resides in facility that provides on-site medical care (e.g., skilled nursing facility)
* Domestic violence screen positive

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2021-02-18 (Actual); Primary Completion 2021-05-07 (Actual); Study Completion 2021-05-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Utah Health, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hung WW, Ross JS, Farber J, Siu AL. Evaluation of the Mobile Acute Care of the Elderly (MACE) service. JAMA Intern Med. 2013 Jun 10;173(11):990-6. doi: 10.1001/jamainternmed.2013.478. PMID 23608775
- [Background] Fong TG, Tulebaev SR, Inouye SK. Delirium in elderly adults: diagnosis, prevention and treatment. Nat Rev Neurol. 2009 Apr;5(4):210-20. doi: 10.1038/nrneurol.2009.24. PMID 19347026
- [Background] 2014 National and State Healthcare-Associated Infections Progress Report.; 2016. http://www.cdc.gov/hai/surveillance/progress-report/index.html. Accessed April 19, 2016.
- [Background] Counsell SR, Holder CM, Liebenauer LL, Palmer RM, Fortinsky RH, Kresevic DM, Quinn LM, Allen KR, Covinsky KE, Landefeld CS. Effects of a multicomponent intervention on functional outcomes and process of care in hospitalized older patients: a randomized controlled trial of Acute Care for Elders (ACE) in a community hospital. J Am Geriatr Soc. 2000 Dec;48(12):1572-81. doi: 10.1111/j.1532-5415.2000.tb03866.x. PMID 11129745
- [Background] Leff B, Burton L, Mader SL, Naughton B, Burl J, Inouye SK, Greenough WB 3rd, Guido S, Langston C, Frick KD, Steinwachs D, Burton JR. Hospital at home: feasibility and outcomes of a program to provide hospital-level care at home for acutely ill older patients. Ann Intern Med. 2005 Dec 6;143(11):798-808. doi: 10.7326/0003-4819-143-11-200512060-00008. PMID 16330791
- [Background] Cryer L, Shannon SB, Van Amsterdam M, Leff B. Costs for 'hospital at home' patients were 19 percent lower, with equal or better outcomes compared to similar inpatients. Health Aff (Millwood). 2012 Jun;31(6):1237-43. doi: 10.1377/hlthaff.2011.1132. PMID 22665835
- [Background] Levine DM, Ouchi K, Blanchfield B, Diamond K, Licurse A, Pu CT, Schnipper JL. Hospital-Level Care at Home for Acutely Ill Adults: a Pilot Randomized Controlled Trial. J Gen Intern Med. 2018 May;33(5):729-736. doi: 10.1007/s11606-018-4307-z. Epub 2018 Feb 6. PMID 29411238
- [Background] Bureau UC. What is Rural America?https://www.census.gov/library/stories/2017/08/rural-america.html. Published 2017. Accessed May 31, 2019.
- [Background] Garcia MC, Rossen LM, Bastian B, Faul M, Dowling NF, Thomas CC, Schieb L, Hong Y, Yoon PW, Iademarco MF. Potentially Excess Deaths from the Five Leading Causes of Death in Metropolitan and Nonmetropolitan Counties - United States, 2010-2017. MMWR Surveill Summ. 2019 Nov 8;68(10):1-11. doi: 10.15585/mmwr.ss6810a1. PMID 31697657
- [Background] Parker K, Horowitz J, Brown A, Fry R, Cohn D, Igielnik R. What Unites and Divides Urban, Suburban and Rural Communities.; 2018. https://www.pewsocialtrends.org/wpcontent/uploads/sites/3/2018/05/Pew-Research-Center-Community-Type-Full-Report-FINAL.pdf. Accessed May 31, 2019
- [Background] Creditor MC. Hazards of hospitalization of the elderly. Ann Intern Med. 1993 Feb 1;118(3):219-23. doi: 10.7326/0003-4819-118-3-199302010-00011. PMID 8417639
- [Background] Joynt KE, Orav EJ, Jha AK. Mortality rates for Medicare beneficiaries admitted to critical access and non-critical access hospitals, 2002-2010. JAMA. 2013 Apr 3;309(13):1379-87. doi: 10.1001/jama.2013.2366. PMID 23549583
- [Background] Joynt KE, Harris Y, Orav EJ, Jha AK. Quality of care and patient outcomes in critical access rural hospitals. JAMA. 2011 Jul 6;306(1):45-52. doi: 10.1001/jama.2011.902. PMID 21730240

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A patient may be considered for Rural home hospital care if they are acutely ill at home, present acutely ill to a clinic or emergency department, or if they are admitted and require additional days of acute care. They must meet inclusion and exclusion criteria and be assessed for eligibility by the rural home hospital physician. Clinicians are any member of the rural home hospital clinical team that will be providing care to rural patients that enroll in the intervention.
Pre-assignment Details: No significant event occurred after participant enrollment
Groups:
- Patients: Patients who received the home hospital intervention. Patients receive hospital-level care in their home, as a substitute to traditional hospital care.
- Clinicians: Clinicians that provide hospital-level care in a patient's home, as a substitute to traditional hospital care.
  Home hospital care: Patients receive hospital-level care in their home.
Period: Overall Study
Arm/Group | Patients | Clinicians
Started | 3 (3 patients were enrolled in this study) | 4 (4 clinicians were enrolled in this study)
Completed | 3 (3 patients were enrolled in this study) | 4 (4 clinicians were enrolled in this study)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The baseline analysis population only includes patients. Baseline characteristics were not collected for clinicians
Groups:
- Patients: Patients receive hospital-level care in their home, as a substitute to traditional hospital care.
  Home hospital care: Patients receive hospital-level care in their home.
- Total: Total of all reporting groups
Arm/Group | Patients | Clinicians | Total
Number analyzed (Participants) | 3 | 0 | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 0 | 1
  >=65 years | 2 | 0 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 77 (12) |  | 77 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 |  | 3
  Male | 0 |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0
  Asian | 0 |  | 0
  Native Hawaiian or Other Pacific Islander | 0 |  | 0
  Black or African American | 0 |  | 0
  White | 3 |  | 3
  More than one race | 0 |  | 0
  Unknown or Not Reported | 0 |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 |  | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients That Completed Their Rural Home Hospitalization
Description: Rural home hospital is when eligible rural patients receive hospital level care at home. This measure includes patients that were hospitalized in rural home hospital for treatment for their acute condition and were discharged from rural home hospital after their treatment was complete. The number in the data table reflects the number of patients that completed their home hospitalization.
Time Frame: Day of admission to day of discharge, estimated 10 days later
Population: Three patients completed a rural home hospitalization. Rural home hospitalized patients were treated for their acute condition in rural home hospital.
Measure: Count of Participants; unit: Participants
Arm/Group | Patients
Number analyzed (Participants) | 3
Participants | 3

2. Secondary Outcome: 3-item Care Transition Measure
Description: This is a hospital level measure of performance that reports the average patient reported quality of preparation for self-care response among adult patients discharged from general acute care hospitals. Data will be collected by a Research Assistant via patient, ( scale of 1 to 12; where 12 indicates highest readiness to transition). The final score is calculated by calculating the sum or responses across the three items ((score Strongly Disagree = 1; Disagree = 2; Agree = 3; Strongly Agree = 4), the number of questions answers are counted, and then the mean response is then calculated (sum divided by count).
Time Frame: Once, within Day of discharge to 7 days later
Population: Rural home hospitalized patients that completed the discharge survey
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Patients
Number analyzed (Participants) | 1
score on a scale | 12 (0)

3. Secondary Outcome: Picker Experience Questionnaire
Description: The Picker Patient Experience Questionnaire is a fifteen item questionnaire covering eight domains including information & education and coordination of care. The questionnaire is used to measure patient experience with in-patient care. The questions have two ("yes" or "no") to four response options ("yes"," no", "I did not need to", or "yes, to some extent"). Neutral answers, such as "I did not need to", and the most positive answer are coded as a "non-problem" (score = 0). The remaining responses are coded as "problems" (score = 1). A problem is defined as any aspect of health care that could be improved upon. Data will be collected by a research assistant via patient. Scale of 1-15, where a higher score indicates better patient experience.
Time Frame: Once, within Day of discharge to 7 days later
Population: Rural home hospitalized patients that completed the discharge survey
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Patients
Number analyzed (Participants) | 1
score on a scale | 13 (0)

4. Secondary Outcome: Global Satisfaction: Scale
Description: Measure of patient experience and satisfaction with care using any number from 0 to 10, where 0 is the worst hospital possible and 10 is the best hospital possible. Data will be collected by a Research Assistant via patient
Time Frame: Once, between Day of discharge to 7 days later
Population: Rural home hospitalized patients that completed the discharge survey
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Patients
Number analyzed (Participants) | 1
score on a scale | 10 (0)

5. Secondary Outcome: Perceived Acceptability of RHH Care
Description: Perceived acceptability will be assessed qualitatively through post-discharge semi-structured interviews with clinicians, patients, and caregivers.The numbers in the data table reflect the number of patients and clinicians that perceived rural home hospital care to be acceptable.
Time Frame: Day of discharge to 30 days later
Population: Only one patient that completed home hospital hospitalization completed a qualitative interview post discharge therefore qualitative data was collected from only one patient. Four clinicians completed qualitative interviews and therefore qualitative data from four clinicians was analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Patients | Clinicians
Number analyzed (Participants) | 1 | 4
Participants | 1 | 4

6. Secondary Outcome: Perceived Safety, Quality of Care, Caregiver Burden
Description: Perceived safety, quality of care, caregiver burden will be assessed qualitatively through one post-discharge semi-structured interview with each participating clinician, patient, and caregiver.
  The numbers in the data table reflect the number of patients and clinicians that perceived that rural home hospital was safe and that the care provided was of high quality.
Time Frame: Day of discharge to 30 days later
Population: One patient that completed home hospital hospitalization completed a qualitative interview post discharge therefore qualitative data was collected from only one patient. Four clinicians completed qualitative interviews
Measure: Count of Participants; unit: Participants
Arm/Group | Patients | Clinicians
Number analyzed (Participants) | 1 | 4
Participants | 1 | 4

7. Secondary Outcome: Number of Rural Home Hospital Patients Escalated to Hospital for Care
Description: If enrolled patient must be discharged from rural home hospital and taken to an acute-care hospital for care. Data to be collected daily by a research assistant via the Registered Nurse or Paramedic
Time Frame: Day of admission to day of discharge, estimated 10 days later
Population: Three patients were enrolled in this study, these patients received the home hospital intervention. Patients receive hospital-level care in their home, as a substitute to traditional hospital care.
Measure: Count of Participants; unit: Participants
Arm/Group | Patients
Number analyzed (Participants) | 3
Participants | 0

8. Secondary Outcome: Number of Patients With an Adverse Event
Description: Adverse events include Fall, Delirium, Potentially preventable Venous Thromboembolism (VTE), New pressure ulcer, Thrombophlebitis at peripheral intravenous line (IV) site. Data to be collected daily by a research assistant via the Registered Nurse or Paramedic
Time Frame: Day of admission to day of discharge, estimated 10 days later
Measure: Count of Participants; unit: Participants
Groups:
- Patients: Patients who received the home hospital intervention
Arm/Group | Patients
Number analyzed (Participants) | 3
Participants | 0

9. Secondary Outcome: Number of Patients With Unplanned Mortality During Admission
Description: Any case of unplanned death among enrolled rural home hospital patient.Data to be collected daily by a research assistant via the Registered Nurse or Paramedic
Time Frame: Day of admission to day of discharge, estimated 10 days later
Measure: Count of Participants; unit: Participants
Arm/Group | Patients
Number analyzed (Participants) | 3
Participants | 0

10. Secondary Outcome: Lab Orders, Number
Description: Number of clinical lab orders. Data to be collected daily by a research assistant via rural home hospital records
Time Frame: Day of admission to day of discharge, estimated 10 days later
Population: Patients that were home hospitalized
Measure: Number; unit: lab orders
Arm/Group | Patients
Number analyzed (Participants) | 3
lab orders | 0

11. Secondary Outcome: Length of Stay
Description: The number of days enrolled patient is admitted to rural home hospital.Data to be collected daily by a research assistant via rural home hospital records.
Time Frame: Day of admission to day of discharge, estimated 10 days later
Population: Patients that were home hospitalized
Measure: Mean (Standard Deviation); unit: number of days
Arm/Group | Patients
Number analyzed (Participants) | 3
number of days | 5.5 (0.57)

12. Secondary Outcome: Unplanned Readmission(s), Number or Patients
Description: Unplanned readmission of patient to hospital 30 days post discharge from rural home hospital. Data to be collected by a research assistant via the patient.
Time Frame: 30-days post-discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Patients
Number analyzed (Participants) | 3
Participants | 0

13. Secondary Outcome: ED Visit(s), Number
Description: Any Emergency Department (ED) visits 30 days post-discharge from rural home hospital. Data to be collected by a research assistant via the patient
Time Frame: 30-days post-discharge
Population: Patients that were home hospitalized
Measure: Number; unit: number of ED visits
Arm/Group | Patients
Number analyzed (Participants) | 3
number of ED visits | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the start of the study through study completion. This was a period of three months in total.
Description: No serious adverse events were reported and there was no risk for all-cause mortality.
Groups:
- Patients: Patients who received the home hospital intervention. Patients receive hospital-level care in their home, as a substitute to traditional hospital care. Adverse events were monitored only for patients.
- Clinicians: Adverse events were not monitored for clinicians.
Arm/Group | Patients | Clinicians
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/0
Other Adverse Events (participants affected / at risk) | 0/3 | 0/0

LIMITATIONS AND CAVEATS:
Our study has limitations.1. We admitted three patients from two rural areas of Utah, limiting generalizability. Second, two out of three patients were lost to follow-up and did not complete a discharge survey or interview. These patients may have had experiences we did not capture.Third, given this was a small proof of concept, the technology systems were not integrated by design.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-20): https://cdn.clinicaltrials.gov/large-docs/80/NCT04531280/Prot_SAP_000.pdf